CLINICAL TRIAL: NCT01105026
Title: Bone Regeneration by Means of a Bioactive Glass Scaffold.
Brief Title: A Clinical Investigation to Evaluate the Healing of Tooth Extraction Sites Filled With BioRestore™
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Trieste (Other)
Collaborators: Inion Oy (Industry)
Responsible Party: Dr. Clozza Emanuele, Division of Dental Sciences and Biomaterials, Department pf Biomedicine, University of Trieste, Trieste, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT-109-CT
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2009-11

CONDITIONS: Alveolar Bone Loss
Keywords: alveolar ridge preservation, bioactive glass, tooth extraction, graft material
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bioactive glass (Experimental)
  Interventions: Device: Alveolar Bone Defect Regeneration Following Tooth Extraction

INTERVENTIONS:
Device: Alveolar Bone Defect Regeneration Following Tooth Extraction — Patients underwent surgery under local anesthesia and minimally invasive periotomy was carried out with a surgical blade. Atraumatic extraction with forceps was performed. The extraction socket was carefully curetted to remove the granulation tissue and was rinsed with a physiologic solution. To evaluate the eligibility of the surgical site, the alveolar walls integrity was checked clinically and by means of extemporaneous peri-apical radiography.
  Then, the socket was filled to the bone margin with Inion BioRestore™ (granules size 1 to 2 millimetres). Finally, single interrupted (5-0) sutures were tightened to promote the stability of grafted particles. Ten days after the surgery, sutures were removed.

SUMMARY:
The aim of this study was to evaluate by histology and MSCT scans during a 7-month period, the efficacy of a bioactive glass (Inion BioRestore™) placed in human extraction sockets in the maintenance of alveolar ridge.

DETAILED DESCRIPTION:
14 subjects in need of implant therapy were enrolled in the study. A total of 32 teeth were extracted and the fresh sockets underwent to ridge preservation procedures using Inion BioRestore™. Two different time points (1 week and 3 months after RPP) MSCT scans for each patient were used as a basis for bone change analysis occurred in the localized grafted alveolar sites. Twenty-two biopsied, representative of intermediate (3-4 months, n=10) and late phase (6-7 months, n=12) of healing, were harvested and histologically analysed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy females or males subjects.
* They did not smoke
* Did not take any medications.

Exclusion Criteria:

* Subjects with less than 18 years of age,
* with current alcohol or drug abuse,
* with systemic/local conditions that would interfere with wound healing or osseointegration
* with a history of chemotherapy and radiotherapy in the head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

REFERENCES:
- [Derived] Clozza E, Biasotto M, Cavalli F, Moimas L, Di Lenarda R. Three-dimensional evaluation of bone changes following ridge preservation procedures. Int J Oral Maxillofac Implants. 2012 Jul-Aug;27(4):770-5. PMID 22848877
- [Derived] Clozza E, Pea M, Cavalli F, Moimas L, Di Lenarda R, Biasotto M. Healing of fresh extraction sockets filled with bioactive glass particles: histological findings in humans. Clin Implant Dent Relat Res. 2014 Feb;16(1):145-53. doi: 10.1111/j.1708-8208.2012.00463.x. Epub 2012 Jun 12. PMID 22691124